CLINICAL TRIAL: NCT04697927
Title: Ascertainment of Epidemiologic Risk Information to Assess Susceptibility to and Severity of SARS-CoV-2 Infection
Brief Title: A Study of Risk Factors for the COVID-19 Virus Infection
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-418
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: COVID-19 Infections in Cancer Patients
Keywords: SARS-CoV-2 infection; Questionnaires; 20-418
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MSK Patients: Patients include those undergoing cancer screening and treatment as well as cancer survivors that received COVID-related care. Both adult and pediatric patients will be included.
  Interventions: Other: Questionnaires
- Household Members (identified by MSK Patient): Individuals over the age of 18 (i.e., individuals currently living in the same household as the MSK enrollee).
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — The epidemiologic questionnaires used in this study are a composite of validated questions from multiple sources. Many of the questions are an expansion of the MSK General Medical Health clinical questionnaire. Validated questions capturing demographics, employment, risk behaviors, family history, as well as, specific research domains including psychosocial, food security, and financial toxicity have already been utilized in other MSK minimal risk studies. The COVID-19 symptom and history tracker questions were largely drawn from the COronavirus Pandemic Epidemiology (COPE) consortium study.

SUMMARY:
The purpose of this study is to collect information that will help the reasearchers learn more about COVID-19 infections in cancer patients, and to find out about the effects of these infections on cancer treatment and outcomes. The research study involves asking people to complete a series of online questionnaires that include questions about their medical history, lifestyle, and risk factors related to the COVID-19 infection. The study will enroll both MSK patients and their household family members.

ELIGIBILITY:
Inclusion Criteria:

MSK Patients

* All individuals who have had at least one point of contact since January 1st 2019 as a patient, including visiting an MSK facility for treatment, clinical evaluation, follow-up or screening, COVID-related screening, or a telehealth visit. Household Members of MSK Patients
* Individuals aged 18 or older
* Currently reside in the same household of MSK patients enrolled onto this protocol
* Have an email account

Exclusion Criteria:

* Impaired decision-making capacity as noted in EHR
* Current MSK employee

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As this is an institution-wide registry, potential research subjects will be identified by the Health Informatics group.
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
develop a comprehensive registry database | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonine Bernstein, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm